CLINICAL TRIAL: NCT01713556
Title: Treatment of PTSD by Reduction of Traumatic Memory Reconsolidation by Propranolol : a Multisite Trial
Acronym: REDUCTRAUMA2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09 106 01
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Post-traumatic Stress Disorder
Keywords: PTSD, Propranolol
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propranolol + reactivation (Experimental): they have a script-driven mental imagery of the traumatic event white drug
  Interventions: Drug: Propranolol; Other: Trauma reactivation
- Placebo + reactivation (Placebo Comparator): They have a script-driven mental imagery of the traumatic event with placebo
  Interventions: Other: Trauma reactivation; Drug: placebo

INTERVENTIONS:
Drug: Propranolol
  Arms: Propranolol + reactivation
Other: Trauma reactivation — Trauma reactivation: script-driven mental imagery of the traumatic event
Drug: placebo
  Arms: Placebo + reactivation

SUMMARY:
The purpose of this study is to test whether propranolol, when given during a re-evocation of a traumatic memory, is capable of reducing subsequent PTSD symptoms associated with that memory.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) develops following an exposure to a life threatening event. One of the characteristic features of PTSD is the recurrence of intrusive memories of an experienced trauma. The persistence of disturbing traumatic memories in PTSD is often explained in terms of a trauma-induced enhancement of memory encoding. Several studies indicate that an increased noradrenergic activity during trauma enhances the encoding of memory. Elevated levels of norepinephrine in the cerebrospinal fluid of individuals with PTSD and the correlation of this elevation with the severity of PTSD symptoms suggest that increased noradrenergic activity is also involved in the maintenance of PTSD symptoms. Reactivation of memory by retrieval also renders the memory labile and susceptible to treatments. This latter process is referred to as memory reconsolidation. Consolidation and reconsolidation both occur within a distinct time window following new learning (in consolidation) and/or retrieval (in reconsolidation). Even well-consolidated old fear memories undergo reconsolidation and may be disrupted by means of pharmacological manipulation. Propranolol may be effective in treating PTSD long after symptoms have been consolidated. Propranolol given after reactivation of the memory of a past traumatic event reduces physiologic responding during subsequent mental imagery of the event.

HYPOTHESE: Subjects with chronic PTSD who receive propranolol before trauma evocation will subsequently show decreased PTSD symptoms, compared to subjects who receive a placebo.

METHOD: 56 participants with chronic PTSD will be recruited for participation. On Week 1, the subjects will complete a standardized measure of PTSD symptoms. Next, 90 minutes after the administration of the study medication (either propranolol or placebo), participants will undergo a script preparation procedure, during which they will disclose details of their traumatic event. Scripts portraying this event will be prepared for subsequent replay.

On Week 2, after the administration of the study medication (either propranolol or placebo), participants will be asked (reading the script) to engaged in a script-driven mental imagery of the traumatic event. Following this procedure, PTSD symptoms will be assessed.

The same procedure will be repeated on Weeks 3, 4, 5 and 6. On Weeks 7 and 18, the standardized measure of PTSD symptoms will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic PTSD
* PTSD CheckList total score >44

Exclusion Criteria:

* Systolic blood pressure < 100 mmHg
* Contraindication to Propranolol
* Previous adverse reaction to a β-blocker
* Use of another β-blocker
* Use of medication that could involve potentially dangerous interactions with propranolol
* Psychotherapy or treatment with any pharmacologic PTSD medication within the 2 weeks prior to inclusion (6 weeks for fluoxetine)
* Female with reproductive potential without reliable means of contraception
* Pregnancy or lactation
* Alcohol or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
PTCD CheckList (PCL) total score. | difference between week 1 (before administration of the study medication) and week 7 (one week after the last intake of study medication)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BIRMES, MD, Principal Investigator — University Hospital, Toulouse
Locations (4):
- France (4):
  - Centre Hospitalier Charles Perrens, Bordeaux
  - Chru Lille, Lille
  - Chu Montpellier, Montpellier
  - CHU Toulouse, Toulouse

REFERENCES:
- [Derived] Roullet P, Vaiva G, Very E, Bourcier A, Yrondi A, Dupuch L, Lamy P, Thalamas C, Jasse L, El Hage W, Birmes P. Traumatic memory reactivation with or without propranolol for PTSD and comorbid MD symptoms: a randomised clinical trial. Neuropsychopharmacology. 2021 Aug;46(9):1643-1649. doi: 10.1038/s41386-021-00984-w. Epub 2021 Feb 21. PMID 33612830